CLINICAL TRIAL: NCT03614598
Title: Impact on Postoperative Pain of Three Single-use Adult Supraglottic Airway Devices in Short General Anesthetic Under Controlled Ventilation
Acronym: DISPOSITIF LAR
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre Hospitalier Universitaire de Nīmes (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: Local/2008/JL- 02; 2008-A00741-54 (Other: ANSM)
Record Dates: First submitted 2018-07-20; First posted 2018-08-03 (Actual); Last update posted 2025-11-17 (Actual); Status verified 2025-11

CONDITIONS: Pharyngolaryngeal Postoperative Pain

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- LMA-UNIQUE™ (Active Comparator)
  Interventions: Procedure: Insertion of LMA-UNIQUE(TM) device
- LMA-SUPREME™ (Active Comparator)
  Interventions: Procedure: Insertion of LMA-SUPREME(TM) device
- I-GEL® (Active Comparator)
  Interventions: Procedure: Insertion of I-GEL(R) device

INTERVENTIONS:
Procedure: Insertion of LMA-UNIQUE(TM) device — LMA-UNIQUE(TM) single-use adult supraglottic airway device inserted during short general anesthesia under controlled ventilation
  Arms: LMA-UNIQUE™
Procedure: Insertion of LMA-SUPREME(TM) device — LMA-SUPREME(TM) single-use adult supraglottic airway device inserted during short general anesthesia under controlled ventilation
  Arms: LMA-SUPREME™
Procedure: Insertion of I-GEL(R) device — I-GEL(R) single-use adult supraglottic airway device inserted during short general anesthesia under controlled ventilation
  Arms: I-GEL®

SUMMARY:
The investigators hypothesize that incidence of pharyngolaryngeal postoperative pain caused by the I-gel and LMA-Suprême devices will be ≤ 5%

ELIGIBILITY:
Inclusion Criteria:

* The patient must have given their free and informed consent and signed the consent form
* The patient must be a member or beneficiary of a health insurance plan
* Adult patients > 18
* ASA score I-III
* Patient scheduled to undergo elective surgery lasting less than two hours under general anaesthetic without tracheal intubation
* The subject is participating in an interventional study, or is in a period of exclusion determined by a previous study
* The subject refuses to sign the consent
* It is impossible to give the subject informed information
* The patient is under safeguard of justice or state guardianship
* The patient is pregnant or breastfeeding
* Emergency surgery
* Sore thoat ≤ 1 month
* Risk of aspiration of gastric contents
* Body mass index (BMI) > 35
* Patients with expected airway difficulties
* Contra-indication for any of the devices (symptomatic hiatal hernias, pathological obesity, poly trauma or serious injury, delayed gastric emptying, use of opiates during fasting)
* Patients who are not fasting for routine and emergency anesthesia
* Trismus, limited mouth opening, abscess or pharyngoperilaryngeal mass

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 546 (Actual)
Dates: Start 2009-04-22 (Actual); Primary Completion 2012-09-05 (Actual); Study Completion 2012-09-06 (Actual)

PRIMARY OUTCOMES:
Incidence of pharyngolaryngeal postoperative pain of the three devices | 24 hours
  Sore throat Y/N

SECONDARY OUTCOMES:
Pharyngolaryngeal postoperative pain between groups | 2 hours
  Sore throat Y/N
Time taken to place device | End of surgery (maximum 2 hours)
  From first attempt at introduction until acceptable exhaled CO2 curve attained (seconds)
Number of attempts needed to place device | End of surgery (maximum 2 hours)
Necessity of altering the size of the device | End of surgery (maximum 2 hours)
  Y/N
Any patient movement during procedure | End of surgery (maximum 2 hours)
  Y/N
Difficulty of insertion | End of surgery (maximum 2 hours)
  5-point scale: very easy-failure
Total leakage pressure of the devices | End of surgery (maximum 2 hours)
  measured directly by the respirator
Ventilatory pressure of the devices | End of surgery (maximum 2 hours)
Device stability during surgery | End of surgery (maximum 2 hours)
  Need to change the management system airways (orotracheal intubation or others) Y/N
Difficulty of device removal | End of surgery (maximum 2 hours)
  4-point scale: very easy-very difficult

CONTACTS AND LOCATIONS:
Overall Officials: Joël L'Hermite, MD, Principal Investigator — CHU Nimes
Locations (1):
- CHU Nimes, Nîmes, France

REFERENCES:
- [Result] L'Hermite J, Dubout E, Bouvet S, Bracoud LH, Cuvillon P, Coussaye JE, Ripart J. Sore throat following three adult supraglottic airway devices: A randomised controlled trial. Eur J Anaesthesiol. 2017 Jul;34(7):417-424. doi: 10.1097/EJA.0000000000000539. PMID 27755181